CLINICAL TRIAL: NCT07326774
Title: Evaluation of the Effect of Ultrasound-Guided Quadro-Iliac Plane Block on Postoperative Analgesia in Patients Undergoing Lumbar Spinal Surgery
Brief Title: Effect of Ultrasound-Guided Quadro-Iliac Plane Block on Postoperative Analgesia After Lumbar Spinal Surgery
Status: Not yet recruiting | Type: Observational
Sponsor: Fatih Sultan Mehmet Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Elif Acar Değer, Dr, Fatih Sultan Mehmet Training and Research Hospital
Other Study IDs: 2025/397
Record Dates: First submitted 2025-12-26; First posted 2026-01-08 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Postoperative Pain; Lumbar Spine Surgery; Postoperative Analgesia
Keywords: Quadro-Iliac Plane Block; QIPB; Ultrasound-Guided Regional Anesthesia; Lumbar Spinal Surgery; Postoperative Analgesia; Patient-Controlled Analgesia
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PCA + QIPB Group: Patients who receive standard postoperative intravenous patient-controlled analgesia (PCA) with tramadol in combination with ultrasound-guided Quadro-Iliac Plane Block (QIPB) as part of routine clinical care following lumbar spinal surgery.
  Interventions: Other: QIPB
- PCA Only Group: Patients who receive standard postoperative intravenous patient-controlled analgesia (PCA) with tramadol alone without the addition of any regional analgesic block following lumbar spinal surgery.

INTERVENTIONS:
Other: QIPB — Quadro-Iliac Plane Block using local anesthetic.
  Groups: PCA + QIPB Group

SUMMARY:
This prospective observational study aims to evaluate the effect of ultrasound-guided Quadro-Iliac Plane Block (QIPB) on postoperative analgesia in patients undergoing lumbar spinal surgery. Lumbar spinal procedures are commonly associated with significant postoperative pain, which may impair early mobilization and increase opioid consumption. In routine clinical practice, QIPB is increasingly used as part of multimodal analgesia to improve pain control and reduce opioid-related adverse effects.

Adult patients scheduled for elective lumbar spinal surgery under general anesthesia will be followed according to routine clinical care. Postoperative analgesia will be managed with intravenous patient-controlled analgesia (PCA) using tramadol, with or without the addition of ultrasound-guided QIPB, based on the preference of the attending anesthesiologist. No intervention or treatment assignment will be performed by the investigators.

Postoperative pain scores at rest and during movement, opioid consumption, need for rescue analgesics, incidence of nausea and vomiting, and patient satisfaction will be recorded during the first 24 hours after surgery. The findings of this study are expected to provide further clinical evidence regarding the effectiveness of QIPB as part of multimodal analgesia in lumbar spinal surgery.

DETAILED DESCRIPTION:
This is a single-center, prospective observational cohort study conducted in patients undergoing elective lumbar spinal surgery under general anesthesia. The study is designed to assess the effects of ultrasound-guided Quadro-Iliac Plane Block (QIPB) on postoperative analgesia when used as part of routine multimodal pain management.

Eligible patients aged 18-65 years with American Society of Anesthesiologists (ASA) physical status I-III and a body mass index below 35 kg/m² will be included after providing written informed consent. All patients will receive standardized general anesthesia and postoperative intravenous patient-controlled analgesia (PCA) with tramadol as part of routine care. The decision to perform QIPB will be made by the attending anesthesiologist according to clinical judgment and routine practice, without any intervention or assignment by the research team.

Ultrasound-guided QIPB, when applied, will be performed bilaterally under sterile conditions in the prone position at the end of surgery. Patients will be observed in two cohorts: those receiving PCA alone and those receiving PCA in combination with QIPB.

Postoperative outcomes will be assessed in the post-anesthesia care unit and at 1, 6, 12, and 24 hours postoperatively. Pain intensity will be evaluated using the Numeric Rating Scale (NRS) at rest and during movement. Secondary outcomes will include total opioid consumption, time to first rescue analgesic requirement, incidence of postoperative nausea and vomiting, sedation level, and patient satisfaction assessed using a 5-point Likert scale at 24 hours. Any block-related complications will also be recorded.

Data will be analyzed using appropriate statistical methods to compare postoperative analgesic outcomes between the two cohorts. This observational study aims to reflect real-world clinical practice and contribute to the growing evidence on the role of QIPB in postoperative pain management after lumbar spinal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 65 years
* American Society of Anesthesiologists (ASA) physical status I-III
* Body mass index (BMI) <35 kg/m²
* Scheduled for elective posterior lumbar spinal instrumentation surgery under general anesthesia

Exclusion Criteria:

* Refusal to participate in the study
* Emergency surgery
* Local infection or hematoma at the block application site
* Previous surgery at the block application site
* Presence of coagulopathy
* Known allergy or toxicity to local anesthetics
* History of hematological, renal, or hepatic disease, or advanced respiratory or cardiac failure
* Chronic analgesic use, chronic alcohol consumption, or substance abuse
* Inability to speak Turkish or presence of language/communication barriers

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients aged 18-65 years with ASA physical status I-III and body mass index <35 kg/m² scheduled for elective posterior lumbar segmental instrumentation surgery under general anesthesia. All participants provide written informed consent prior to enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain Intensity | Within the first 24 hours after surgery
  Postoperative pain intensity assessed using the Numeric Rating Scale (NRS), where 0 indicates no pain and 10 indicates the worst imaginable pain.

SECONDARY OUTCOMES:
Total Opioid Consumption | Within the first 24 hours after surgery
  Total amount of tramadol consumption administered via intravenous patient-controlled analgesia during the first 24 hours postoperatively.
Requirement for Rescue Analgesia | Within the first 24 hours after surgery
  Need for additional rescue analgesic medication during the first 24 hours postoperatively.
Postoperative Nausea and Vomiting | Within the first 24 hours after surgery
  Incidence of postoperative nausea and vomiting during the first 24 hours after surgery.
Patient Satisfaction With Pain Management | 24 hours after surgery
  Patient satisfaction with postoperative pain management was assessed at 24 hours after surgery using a 5-point Likert Satisfaction Scale (range: 1-5), where 1 = "not satisfied at all," 2 = "not satisfied," 3 = "neutral," 4 = "satisfied," and 5 = "very satisfied," with higher scores indicating greater patient satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Oznur Demiroluk, Assoc. Prof., Principal Investigator — Fatih Sultan Mehmet Training and Research Hospital, Istanbul, Türkiye
Locations (1):
- Fatih Sultan Mehmet Training and Research Hospital, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared, as data sharing was not planned at the time of study design and is not included in the ethical approval.